CLINICAL TRIAL: NCT01262209
Title: Clinical Effectiveness of Low Vision Rehabilitation in Glaucoma Patients With Moderate or Severe Vision Loss
Brief Title: Clinical Effectiveness of Low Vision Rehabilitation in Glaucoma Patients
Acronym: LOVIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Cindy Hutnik, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R-10-481; 17356 (Other: REB)
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Glaucoma
Keywords: Vision loss; Chronic glaucoma; Low vision rehabilitation
MeSH Terms: conditions — Glaucoma; Vision Disorders | interventions — Telescopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low Vision Aids (Experimental): All patients will receive:
  1. A low vision examination:
     1. Low vision refraction
     2. Distance best corrected visual acuity
     3. Near best corrected visual acuity
     4. Contrast Sensitivity
     5. Quality of life questionnaire
  2. Low vision therapy: to teach strategies for more effective use of remaining vision and use of low-vision devices
  3. Prescribed low vision devices including binocular telescope (2.1x or 3.5x), monocular telescope, 6x telemicroscopes, microscopes, magnifiers, portable CCTV and absorptive filters.
  Interventions: Device: portable CCTV; Device: Telescopes, telemicroscopes and microscopes; Device: Absorptive filters

INTERVENTIONS:
Device: portable CCTV — This is a small handheld mini screen intended to improve reading.
Device: Telescopes, telemicroscopes and microscopes — These are either worn like glasses, or held in one's hand and are intended to improve distance vision (like details of a hockey game), intermediate vision (like reading a sign), or 'up-close' vision (like reading small print).
Device: Absorptive filters — These are worn like glasses, and have tinted colour lenses. They are intended to improve contrast sensitivity, or being able to tell light from dark (like reading gray letters on a white background).

SUMMARY:
Our team is interested in what can be done to improve the functioning of patients who suffer from glaucoma, a chronic and irreversible eye disease. Patients with vision loss as a result of this disease may feel like they have been 'given up on', or lost to our medical system when no further interventions can be offered to treat their eye disease. It is our intent to investigate what alternatives we can provide our patients, instead of simply saying, 'nothing more can be done'. We have learned from studies done on other chronic eye diseases, like age related macular degeneration, that low vision rehabilitation can improve visual function.

What exactly is low vision? It can involve a loss of visual acuity, making activities such as reading or writing a challenge; it can involve loss of contrast sensitivity, making shapes and edges hard to discern, like those of a stair edge, or person's face. It could also involve a loss of peripheral, or side vision which is a symptom common to most glaucoma patients. Whatever the cause of low vision, doing day-to-day activities can become increasingly difficult, and many suffer from a loss of their independence and may even become depressed. Low vision rehabilitation involves helping patients to use their remaining vision in optimal, and sometimes even new, ways. This involves an assessment of a person's baseline vision, and an idea of what their needs are. Patients are then given low vision aids (such as magnifiers, telescopes, video screens which magnify images, and other tools) as well as instructions and support for adapting to living and functioning with altered vision.

Although there currently exists no cure for glaucoma, and we are certainly not promising a reversal of the damage done to the eyes from this chronic disease, we do believe that these types of rehabilitation services may offer some hope and potential visual benefit to patients living with vision loss. Our hypothesis is that the use of state-of-the-art low vision aids in patients with advanced glaucomatous visual loss will provide an improvement in visual tasks and thereby an improvement in quality of life.

DETAILED DESCRIPTION:
Visual impairment, including both low vision and blindness, ranks among the ten most prevalent causes of disability in North America (1). Leading causes of low vision are diseases also associated with an aging population, including age related macular degeneration (ARMD), glaucoma, diabetic retinopathy and optic neuropathies (1). Of these, irreversible vision loss is most commonly caused by ARMD and glaucoma, diseases for which there exists no cure (2). Quality of life and functional ability are negatively impacted by vision loss and blindness (2). Loss of visual ability impairs both mental and physical functioning, limiting activities of daily living (ADL) (eating, dressing, reading, writing, mobilizing, interpersonal communication etc.) (3). Impedance on basic functioning secondary to visual impairment can lead to loss of independence, low self-esteem or depression (3). When pharmacological or surgical interventions prove futile in advanced vision loss, low vision rehabilitation may be the only option for regaining lost function in patients. The goal of low vision rehabilitation is to not restore lost vision but rather utilize the remaining vision to its fullest potential thus enabling patients to reclaim their ADL and thereby their independence.

Our study is based on the Veterans Affairs Low Vision Intervention Trial (LOVIT), a randomized controlled trial conducted by Stelmack et al (4-6). Their goal was to evaluate the efficacy of an outpatient low vision rehabilitation program for patients with moderate to severe vision loss secondary to age related macular degeneration (ARMD). Their intervention was effective in improving all aspects of visual function when compared with the control group. There is very little evidence to support the use of low vision rehabilitation in patients with chronic, irreversible visual loss secondary to glaucoma, and currently no randomized trials have been done. Because the pattern of visual loss is different in ARMD and glaucoma, it is not possible to extrapolate the ARMD data beyond the ARMD cohort. Yet, the ARMD experience has established a proof of principal that can be used in the glaucoma protocol design In patients with advanced glaucomatous optic neuropathy, functional loss often begins with mobility and difficulty ambulating (7). In one study, patients with visual field loss secondary to their glaucoma showed a diminished traffic gap judgement when crossing the street, which lead to an increased risk of harm. As a whole, the group made 23% more errors in identifying a gap as crossable when it was too short to be made safely (7). Another researcher found that 25% of patients with visual field loss in both eyes reported a moderate to severe restriction in their mobility activities overall. In another study, field loss secondary to glaucoma lead to a lower vision-related quality of life score. When examined collectively, these reports and others suggest that those with reduced visual fields and glaucoma experience more falls, more motor vehicle accidents, greater overall difficulty with mobility activities and an overall decreased quality of living (7). Visual acuity can vary over a wide range among patients with moderate to severe glaucoma, but overall, central vision reduction occurs late in the disease. Some studies do show mild central and diffuse reduction in fields in the early stages of glaucoma. As the visual fields and visual acuity decline, patients often note difficulty with glare sensitivity, leaving response times to light and dark adaptations hindered. In summary, the problems most often experienced by patients with advanced glaucoma are related to ambulation, reading, distance spotting and glare. Low vision rehabilitation aims to maximize independence in patients' daily lives by addressing these difficulties.

It would be difficult to argue that low vision aids and rehabilitation in patients with visual loss do not have a positive impact on both patients and their families; however there exists little in the way of randomized controlled clinical trials which evaluate efficacy of outpatient low vision rehabilitation and interdisciplinary strategies to deliver such services. Given the existing shortage of inpatient resources and the staff required to manage such patients, an outpatient program could deemed more cost effective and practical in our limited health care system. Moreover, most available data on the subject focuses on rehabilitation in patients with ARMD. There is very little to support the use of low vision rehabilitation in patients with chronic, irreversible visual loss secondary to glaucoma. As our population ages, we can expect with certainty an increase in the prevalence of visual loss secondary to glaucoma, beginning in the next ten years (12). An evaluation of the efficacy of strategies to address 'untreatable' vision loss, such as those patients with 'end of the line' glaucoma, would be of great significance as we see glaucoma and its devastating effects on vision and subsequently on quality of life increase greatly in the near future. Evidence based models of outpatient low vision rehabilitation programs are needed to support the implementation and delivery of such services for patients suffering from moderate to severe glaucoma, and its devastating impact on daily functioning.

References

1. US Department of Health and Human Services. Vision research a national plan: 1999-2003; NIH Publication No. 98-4120. National Eye Institute, Bethesda MD, 1998: 117-30
2. Evans K, Law S, Walt J, Buchholz P, Hansen J. The quality of life impact of peripheral versus central vision loss with a focus on glaucoma versus age-related macular degeneration. Clinical Ophthalmology 2009:3 433-445
3. Department of Veterans Affairs. Veterans Health Administration, Blind Rehabilitation Service. Coordinated Services for Blinded Veterans IB 11-59 (revised) P87250. Department of Veterans Affairs, Washington DC, 1996.
4. Stelmack JA, Tang XC, Reda DJ, Moran D, Rinne S, Mancil RM, Cummings R, Mancil G, Stroupe K, Ellis N, Massof RW. The Veterans Affairs Low Vision Intervention Trial (LOVIT): design and methodology. Clin Trials. 2007;4(6):650-60.
5. Stelmack JA, Tang XC, Reda DJ, Rinne S, Mancil RM, Massof RW. Outcomes of the Veteran Affairs Low Vision Intervention Trial (LOVIT)
6. Stelmack JA, Moran D, Dean D, Massof RW. Short and long-term effects of an intensive inpatient vision rehabilitation program. Arch Phys Med Rehabil 2007; 88:691-5.
7. Robinson, S. (2010). Chapter 31: Advanced Glaucoma and Low Vision: Evaluation and Treatment. In Schacknow, P.N. and Samples, J.R. (Eds.), The Glaucoma Book: A Practical, Evidence-Based Approach to Patient Care. (pp. 351-353). New York: Springer.
8. Stelmack J, Szlyk J, Stelmack T, et al. Use of Rasch person item map in exploratory data analysis: a clinical perspective. J Rehabil Res Dev 2004; 41: 233-42.
9. Szlyk JP, Stelmack J, Massof RW, et al. Performance of the Veterans Affairs Low Vision Visual Functioning Questionnaire. J Vis Impair Blind 2004; 98: 261-75.
10. Stelmack JA, Szlyk JP, Stelmack TR, et al. Psychometric properties of the Veterans Affairs Low-Vision Visual Functioning Questionnaire. Invest Ophthalmol Vis Sci 2004; 45: 3919-28.
11. Stelmack JA, Szlyk JP, Stelmack TR, et al. Measuring outcomes of low vision rehabilitation with the Veterans Affairs Low Vision Visual Functioning Questionnaire (VALV VFQ-48). Invest Ophthalmol Vis Sci 2006; 47: 3253-61.
12. Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7.

ELIGIBILITY:
Inclusion Criteria:

1. Primary or secondary open angle glaucoma that has been stable for at least 12 months
2. Presenting best corrected visual acuity (in the better seeing eye), measured at the screening visit, better than 20/400 but worse than 20/100 as a result of primary or secondary glaucoma.
3. No surgical or laser procedures in the last 6 months
4. The minimum number of degrees of central visual field (30-2 or 24-2 SITA threshold) should be no less than 20 degrees

Exclusion Criteria:

1. Has no access to telephone
2. Is unable to speak English
3. Has previously received comprehensive low vision services
4. Has English literacy screening less than 5th grade level (Dolch Basic Sight Words List)
5. Has history of stroke with aphasia
6. Has other health condition that would preclude follow-up (e.g., significant malignancy or life-threatening disease)
7. Is unable or unwilling to attend clinic visits required for the study
8. Has severe hearing impairment that interferes with participation in telephone questionnaire
9. Reports significant loss of vision since last eye exam
10. Has macular degeneration, vitreous hemorrhage, serous or hemorrhagic detachment of the macula, clinically significant macular edema or cystoid macular edema that is likely to result in further loss or improvement in vision after treatment in better-seeing eye
11. Planned cataract extraction within the next six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Visual reading ability and visual mobility. | 2 weeks
  The primary outcome measure will be visual reading ability and visual mobility.

SECONDARY OUTCOMES:
Other visual ability domains. | 2 weeks
  Mean changes in other visual ability domains (overall ability, visual information processing and visual motor skills) on the VA LV VFQ-48 from baseline to two weeks are the secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy ML Hutnik, Bsc(Hon), MD, PhD, FRCSC, Principal Investigator — Ivey Eye Institute
Locations (1):
- Ivey Eye Institute, London, Ontario, Canada